CLINICAL TRIAL: NCT00087672
Title: Phase II Study of CC-5013 in Myelofibrosis
Brief Title: A Phase II Study of CC-5013 in Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0648
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Philadelphia negative myeloproliferative disorder; CC-5013; Lenalidomide; Revlimid; Antiangiogenesis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-5013 (Experimental)
  Interventions: Drug: CC-5013

INTERVENTIONS:
Drug: CC-5013 — 10 mg orally (2 capsules) daily
  Other Names: lenalidomide; Revlimid

SUMMARY:
The goal of this clinical research study is to learn if CC-5013 (lenalidomide) can help to control myelofibrosis. The safety of lenalidomide in the treatment of myelofibrosis will also be studied.

DETAILED DESCRIPTION:
Lenalidomide blocks the activity of a substance in the blood called tumor necrosis factor alpha. Tumor necrosis factor alpha is a substance that is believed to prevent new blood cells from forming in the bone marrow. Lenalidomide is also believed to help the body's immune system fight diseases.

Before treatment starts, you will have a complete physical exam, including blood (about 3 teaspoonfuls) and urine tests. A bone marrow sample will be taken. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. An ECG (test to measure the electrical activity of the heart) may be performed.

Women who are able to have children must have a negative pregnancy test [blood (about 1 teaspoon) or urine]. These pregnancy tests must occur within 10 - 14 days and again within 24 hours before the start of lenalidomide. Women who are able to have children with regular or no menstruation must have a pregnancy test weekly for the first 28 days and then every 28 days while on therapy (including breaks in therapy); when they stop taking lenalidomide and at Day 28 after the last dose of lenalidomide. Females with irregular menstruation must have a pregnancy test weekly for the first 28 days and then every 14 days while on therapy (including breaks in therapy), when they stop taking lenalidomide and at Day 14 and Day 28 after the last dose of lenalidomide.

You are considered to be a woman who is able to have children if you are a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

You will take 2 lenalidomide capsules by mouth daily. You should swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

If your platelet count is less than 100,000 at the time of study enrollment, the dose will be one capsule daily. The dose may be decreased depending on side effects. The dose may be increased if needed to better control the disease. This will be decided cycle by cycle.

During treatment, you will give blood samples (about 1 tablespoon each) about every week. The tests may be repeated more frequently to check for side effects. You will need to return to M. D. Anderson monthly for the first 3 months, then at least every 3 months afterwards (while on the study) in order to be evaluated for response and tolerance to lenalidomide. Only one 28-day cycle of lenalidomide may be given to you for each cycle per month.

You may continue to receive this therapy as long as there are no severe side effects or worsening of the disease. You will be asked to keep diaries documenting when you take the capsules. You will also need to return empty medication bottles at each visit. If you have had 4 to 6 months of treatment without any evidence of benefit, you may be taken off the study.

This is an investigational study. Lenalidomide is a new drug related to the drug called thalidomide. Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions. In this case it is considered investigational. Up to 41 participants may take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelofibrosis or Philadelphia negative myeloproliferative disorder with myelofibrosis requiring therapy.
* Disease-free of prior malignancies for greater than or equal to 2 years with exception of basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3.
* Total bilirubin less than or equal to 3.0 mg/dL (unless due to tumor) and serum creatinine less than or equal to 3.0 mg/dL (unless due to tumor).
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
* continued from above.....Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* continued from above.....† A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Signed informed consent.

Exclusion Criteria:

* Use of any other experimental drug or therapy within 28 days of therapy, except in cases with rapidly progressive disease and/or recovery from all toxicity from previous therapy (does not apply to growth factors).
* Platelet count less than 30,000.
* Known prior clinically relevant hypersensitivity reaction or desquamating rash with thalidomide.
* Prior therapy with CC-5013.
* Pregnancy, suspected pregnancy or breast feeding females.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Website for The University of Texas M.D. Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 7/8/04 to 2/27/09. All patients registered at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: The maximum accrual of 41 was met.
Groups:
- CC-5013: 10 mg orally daily
Period: Overall Study
Arm/Group | CC-5013
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CC-5013
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 22
Age Continuous [Median (Full Range); unit: years] | 66 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of CC-5013 in Myelofibrosis
Description: Response evaluation, sustained for 2 weeks: Complete Remission (Neutrophil count between 1 to 10 x 10^9/L without peripheral blasts in blood or bone marrow); Partial Hematologic Response/Partial Remission (Increase in neutrophil by 50% + above 10^9/L for neutropenia); Hematologic Improvement (increase in Neutrophil count, hemoglobin, platelet count or reduction in blood/marrow blasts) or No Response.
  If nine or < patients respond to therapy (response other than 'No Response'), therapy declared ineffective. However, if 11 or > patients respond to therapy, therapy considered efficacious.
Time Frame: 3 - 4 Months for all patients; 24 months for responders
Population: Intention to treat: After a total of 41 patients were enrolled in study, nine or more patients responded to the therapy, therapy declared effective.
Measure: Number; unit: Participants
Arm/Group | CC-5013
Number analyzed (Participants) | 41
Participants
  Complete Remission | 7
  Partial Remission | 9
  Hematologic Improvement | 12
  No Response | 9

ADVERSE EVENTS:
Time Frame: 1 year and 2 months.
Arm/Group | CC-5013
Serious Adverse Events (participants affected / at risk) | 15/41
Other Adverse Events (participants affected / at risk) | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CC-5013 (N=41)
Neutropenic fever (General disorders) | 1 (1) — Unrelated to study drug.
Nausea (Gastrointestinal disorders) | 1 (1) — Unrelated to study drug.
Vomiting (Gastrointestinal disorders) | 1 (3) — Unrelated to study drug.
Pain (General disorders) | 2 (3) — Unrelated to study drug.
Infection (Infections and infestations) | 1 (1) — Unrelated to study drug.
Pneumonia (Infections and infestations) | 2 (2) — Unrelated to study drug
Disease Progression (General disorders) | 1 (1) — Unrelated to study drug.
Infection with neutropenia (Infections and infestations) | 2 (2) — Unrelated to study drug.
Hemorrhage CNS (Vascular disorders) | 1 (1) — Unrelated to study drug.
Death (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (2)
Infection with unknown Absolute neutrophil count (Infections and infestations) | 3 (3)
Edema (Cardiac disorders) | 1 (1) — Unrelated to study drug.
Tachycardia (Cardiac disorders) | 1 (1) — Unrelated to study drug.
Obstruction Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Unrelated to study drug.
Syncope, sensory neuropathy (Nervous system disorders) | 1 (1) — Unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CC-5013 (N=41)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hypomagnesemia (Blood and lymphatic system disorders) | 3 (4)
Infection (Infections and infestations) | 2 (3)
Metabolic/Laboratory (other) (Blood and lymphatic system disorders) | 6 (6)
muscle cramps (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (8)
Neuropathy Sensory (Nervous system disorders) | 6 (6)
Neutrophils (ANC/AGC) (Infections and infestations) | 14 (14) — ANC/AGC = Absolute Neutrophil Count/Absolute Granulocyte Count
pain (headache) (General disorders) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 11 (11)
pruritis (Skin and subcutaneous tissue disorders) | 12 (13)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 16 (21)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No